CLINICAL TRIAL: NCT04516967
Title: Randomized, Double-blind, Placebo-controlled Study With Open-label Extension Phase to Evaluate the Efficacy and Safety of Avatrombopag for the Treatment of Thrombocytopenia in Pediatric Subjects With Immune Thrombocytopenia for ≥6 Months
Brief Title: Avatrombopag for the Treatment of Thrombocytopenia in Pediatric Subjects With Immune Thrombocytopenia for ≥6 Months
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sobi, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVA-PED-301
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Immune Thrombocytopenia
Keywords: ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — avatrombopag

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Experimental: Avatrombopag Double Blind (Experimental): Study is 3:1 randomization ratio (avatrombopag to placebo). Investigational product administered orally once daily for 12 weeks
  Interventions: Drug: Avatrombopag
- Placebo Comparator:Placebo Double Blind (Placebo Comparator): Study is 3:1 randomization ratio (avatrombopag to placebo). Investigational product administered orally once daily for 12 weeks
  Interventions: Drug: Placebo
- Avatrombopag Open Label Extension (Experimental): Investigational product administered orally for up to 2 years.
  Interventions: Drug: Avatrombopag

INTERVENTIONS:
Drug: Avatrombopag — Oral avatrombopag tablet or sprinkle capsule
  Other Names: Doptelet
  Arms: Avatrombopag Open Label Extension; Experimental: Avatrombopag Double Blind
Drug: Placebo — Placebo comparator tablet or sprinkle capsule
  Arms: Placebo Comparator:Placebo Double Blind

SUMMARY:
A Phase 3b Study to Evaluate the Efficacy and Safety of Avatrombopag for the Treatment of Thrombocytopenia in Pediatric Subjects with Immune Thrombocytopenia for ≥6 Months

DETAILED DESCRIPTION:
Subjects will be randomized in to blinded therapy of avatrombopag or placebo in a 3:1 ratio for a period of 12 weeks. Subjects who complete the 12 week treatment period and are eligible may continue to the open label extension phase which will last 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants ≥1 and <18 years of age at Screening and Baseline with a diagnosis of primary ITP for ≥6 months duration and has had an insufficient response to a previous treatment, in the opinion of the Investigator.
* Participant has an average of 2 platelet counts <30×10^9/L with no single count >35×10^9/L in the screening period

Exclusion Criteria:

* Participants must not have a known history of secondary ITP, any history of arterial or venous thrombosis, including partial or complete thrombosis, known inherited thrombocytopenia, a history of myelodysplastic syndrome (MDS) or known history of congenital heart abnormalities or arrhythmias.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2025-10-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (62):
- United States (21):
  - Site 112, Phoenix, Arizona
  - Site 103, Long Beach, California
  - Site 119, Orange, California
  - Site 109, Sacramento, California
  - Site 101, San Francisco, California
  - Site 111, Aurora, Colorado
  - Site 120, Wilmington, Delaware
  - Site 117, Gainesville, Florida
  - Site 116, Atlanta, Georgia
  - Site 107, Peoria, Illinois
  - Site 104, Boston, Massachusetts
  - Site 105, Minneapolis, Minnesota
  - Site 114, Jackson, Mississippi
  - Site 102, Las Vegas, Nevada
  - Site 108, Morristown, New Jersey
  - Site 118, Charlotte, North Carolina
  - Site 113, Durham, North Carolina
  - Site 106, Columbus, Ohio
  - Site 121, Philadelphia, Pennsylvania
  - Site 110, Providence, Rhode Island
  - Site 115, Houston, Texas
- France (2):
  - Site 201, Toulouse, Occitanie
  - Site 202, Paris, Île-de-France Region
- Germany (4):
  - Site 301, Freiburg im Breisgau, Baden-Wurttemberg
  - Site 303, Kiel, Schleswig-Holstein
  - Site 304, Berlin
  - Site 302, Hamburg
- Hungary (3):
  - Site 801, Budapest
  - Site 802, Miskolc
  - Site 803, Pécs
- Poland (5):
  - Site 502, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Site 503, Warsaw, Masovian Voivodeship
  - Site 505, Zabrze, Silesian Voivodeship
  - Site 501, Olsztyn, Warmian-Masurian Voivodeship
  - Site 504, Lodz, Łódź Voivodeship
- Russia (7):
  - Site 907, Chelyabinsk
  - Site 904, Moscow
  - Site 906, Moscow
  - Site 901, Moscow
  - Site 902, Nizhny Novgorod
  - Site 905, Saint Petersburg
  - Site 903, Volgograd
- Turkey (Türkiye) (10):
  - Site 701, Adana
  - Site 704, Ankara
  - Site 706, Antalya
  - Site 702, Antalya
  - Site 705, Denizli
  - Site 709, Istanbul
  - Site 710, Istanbul
  - Site 703, Istanbul
  - Site 707, Izmir
  - Site 708, Mersin
- Ukraine (2):
  - Site 954, Kharkiv, Kharkivs’ka Oblast’
  - Site 952, Vinnytsia
- United Kingdom (8):
  - Site 405, Birmingham, England
  - Site 408, Liverpool, England
  - Site 403, London, England
  - Site 410, London, England
  - Site 407, London, England
  - Site 402, Manchester, England
  - Site 401, Sheffield, England
  - Site 406, Cardiff, Wales

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grace RF, Leblebisatan G, Aydinok Y, Unal S, Grainger JD, Zhang J, Smallwood L, de Leon E, Jamieson BD; AVA-PED-301 Study Group. Avatrombopag for the treatment of children and adolescents with immune thrombocytopenia (AVA-PED-301): a multicentre, randomised, double-blind, placebo-controlled, phase 3b study. Lancet Haematol. 2025 Jul;12(7):e494-e504. doi: 10.1016/S2352-3026(25)00107-3. Epub 2025 May 23. PMID 40418942

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Open label extension optional and not all subjects entered this phase. 73 of 75 entered this phase and 2 dropped out after the core phase.
Groups:
- Avatrombopag Open Label Extension: Subjects receive investigational drug up to 2 years.
Period: Core Phase
Arm/Group | Experimental: Avatrombopag Double Blind | Placebo Comparator:Placebo Double Blind | Avatrombopag Open Label Extension
Started | 54 | 21 | 0
Completed | 44 | 1 | 0
Not Completed | 10 | 20 | 0
Not completed — Adverse Event | 2 | 1 | 0
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Lack of Efficacy | 7 | 18 | 0
Period: Extension Phase
Arm/Group | Experimental: Avatrombopag Double Blind | Placebo Comparator:Placebo Double Blind | Avatrombopag Open Label Extension
Started | 0 | 0 | 73
Completed | 0 | 0 | 4
Not Completed | 0 | 0 | 69

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Avatrombopag: Study is 3:1 randomization ratio (avatrombopag to placebo). Investigational product administered orally once daily for 12 weeks
  Avatrombopag: Oral avatrombopag tablet or sprinkle capsule
- Placebo Comparator:Placebo: Study is 3:1 randomization ratio (avatrombopag to placebo). Investigational product administered orally once daily for 12 weeks
  Placebo: Placebo comparator tablet or sprinkle capsule
- Total: Total of all reporting groups
Arm/Group | Experimental: Avatrombopag | Placebo Comparator:Placebo | Total
Number analyzed (Participants) | 54 | 21 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.9 (4.36) | 9.9 (4.13) | 9.2 (4.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 12 | 36
  Male | 30 | 9 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 50 | 15 | 65
  Unknown or Not Reported | 1 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 48 | 15 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  Turkey | 20 | 9 | 29
  Hungary | 4 | 1 | 5
  United States | 8 | 5 | 13
  Ukraine | 2 | 0 | 2
  Poland | 3 | 1 | 4
  United Kingdom | 11 | 2 | 13
  France | 0 | 1 | 1
  Germany | 2 | 1 | 3
  Russia | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Durable Platelet Response
Description: The proportion of subjects achieving at least 6 out of 8 weekly platelet counts ≥50×10^9/L during the last 8 weeks of the 12 week Treatment Period in the Core Phase, in the absence of rescue medication
Time Frame: Last 8 weeks of 12 week treatment regimen
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Avatrombopag | Placebo Comparator:Placebo
Number analyzed (Participants) | 54 | 21
Participants | 15 | 0
Statistical Analysis 1: Comparison: Experimental: Avatrombopag vs Placebo Comparator:Placebo; Test type: Superiority; p = 0.0077, Fisher Exact

2. Primary Outcome: Alternative Primary: Platelet Response
Description: The proportion of subjects for whom at least 2 consecutive platelet assessments are ≥50×10^9/L over the 12 weeks of treatment in the Core Phase in the absence of rescue medication.
Time Frame: 12 weeks of treatment
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Avatrombopag | Placebo Comparator:Placebo
Number analyzed (Participants) | 54 | 21
Participants | 44 | 0
Statistical Analysis 1: Comparison: Experimental: Avatrombopag vs Placebo Comparator:Placebo; Test type: Superiority; p < 0.0001, Fisher Exact

3. Secondary Outcome: Percentage of Weeks Platelet Count ≥50×10^9/L
Description: The percentage of weeks subjects have a platelet count ≥50×10^9/L during 12 weeks of treatment in the Core Phase, in the absence of rescue therapy.
Time Frame: 12 weeks of treatment
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: percentage of weeks
Arm/Group | Experimental: Avatrombopag | Placebo Comparator:Placebo
Number analyzed (Participants) | 54 | 21
percentage of weeks | 48.9 (25.22) | 1.2 (3.92)
Statistical Analysis 1: Comparison: Experimental: Avatrombopag vs Placebo Comparator:Placebo; Test type: Superiority; p < 0.0001, t-test, 2 sided

4. Secondary Outcome: Platelet Response at Day 8
Description: The proportion of subjects with a platelet count ≥50×10^9/L at day 8, in the absence of rescue therapy.
Time Frame: Day 8
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Avatrombopag | Placebo Comparator:Placebo
Number analyzed (Participants) | 54 | 21
Participants | 30 | 0
Statistical Analysis 1: Comparison: Experimental: Avatrombopag vs Placebo Comparator:Placebo; Test type: Superiority; p < 0.0001, Fisher Exact

5. Secondary Outcome: Percentage of Weeks Platelet Count Between ≥50×10^9/L and ≤150×10^9/L
Description: The percentage of weeks subjects have a platelet count between ≥50×10^9/L and ≤150×10^9/L, during 12 weeks of treatment in the Core Phase, in the absence of rescue therapy.
Time Frame: 12 weeks of treatment
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: percentage of weeks
Arm/Group | Experimental: Avatrombopag | Placebo Comparator:Placebo
Number analyzed (Participants) | 54 | 21
percentage of weeks | 29.2 (19.64) | 1.2 (3.92)
Statistical Analysis 1: Comparison: Experimental: Avatrombopag vs Placebo Comparator:Placebo; Test type: Superiority; p < 0.0001, t-test, 2 sided

6. Secondary Outcome: Rescue Medications
Description: The proportion of subjects who require rescue medications during 12 weeks of treatment in the Core Phase of the study.
Time Frame: 12 weeks of treatment
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Avatrombopag | Placebo Comparator:Placebo
Number analyzed (Participants) | 54 | 21
Participants | 4 | 9
Statistical Analysis 1: Comparison: Experimental: Avatrombopag vs Placebo Comparator:Placebo; Test type: Superiority; p = 0.0008, Fisher Exact

7. Secondary Outcome: Incidence of Any Bleeding Event (WHO Grade 1-4)
Description: Overall incidence of bleeding events associated with ITP measured using the WHO Bleeding Scale (Grade 1-4).
Time Frame: 12 weeks of treatment
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Avatrombopag | Placebo Comparator:Placebo
Number analyzed (Participants) | 54 | 21
Participants | 45 | 19
Statistical Analysis 1: Comparison: Experimental: Avatrombopag vs Placebo Comparator:Placebo; Test type: Superiority; p = 0.7175, Fisher Exact

ADVERSE EVENTS:
Time Frame: Up to 12 weeks (Core Phase) and up to 2 years (ongoing Extension Phase)
Groups:
- Ongoing Open Label Extension Phase: All subjects receive investigational drug for up to 2 years.
Arm/Group | Experimental: Avatrombopag | Placebo Comparator:Placebo | Ongoing Open Label Extension Phase
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/21 | 0/73
Serious Adverse Events (participants affected / at risk) | 5/54 | 1/21 | 16/73
Other Adverse Events (participants affected / at risk) | 50/54 | 16/21 | 62/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Avatrombopag (N=54) | Placebo Comparator:Placebo (N=21) | Ongoing Open Label Extension Phase (N=73)
Immune Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Mouth Haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Oral Purpura (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (5)
Skin Haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Aplastic Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Bone Marrow Disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Bone Marrow Reticulin fibrosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (7)
Dental Caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mucosal Haemorrhage (General disorders) | 0 (0) | 0 (0) | 2 (3)
Hypogammaglobulinaemia (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Abdominal Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Avatrombopag (N=54) | Placebo Comparator:Placebo (N=21) | Ongoing Open Label Extension Phase (N=73)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 0 (0) | 8 (11)
Vomiting (Gastrointestinal disorders) | 4 (6) | 0 (0) | 4 (10)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 4 (12)
Gingival Bleeding (Gastrointestinal disorders) | 2 (2) | 2 (3) | 2 (2)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 9 (9) | 0 (0) | 13 (17)
Upper Respiratory Tract Infection (Infections and infestations) | 6 (6) | 2 (2) | 22 (36)
COVID 19 (Infections and infestations) | 4 (4) | 1 (1) | 3 (4)
Nasopharyngitis (Infections and infestations) | 4 (5) | 0 (0) | 11 (13)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 3 (5) | 0 (0) | 5 (11)
Contusion (Injury, poisoning and procedural complications) | 3 (7) | 1 (1) | 4 (8)
Arthralagia (Musculoskeletal and connective tissue disorders) | 4 (6) | 0 (0) | 3 (6)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 10 (22) | 4 (4) | 10 (32)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 (30) | 4 (9) | 13 (89)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 0 (0) | 13 (27)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0) | 10 (13)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 6 (7)
Petechiae (Skin and subcutaneous tissue disorders) | 14 (20) | 6 (6) | 8 (11)
Ecchymosis (Skin and subcutaneous tissue disorders) | 10 (19) | 1 (1) | 5 (13)
Haematoma (Vascular disorders) | 3 (3) | 3 (6) | 4 (4)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 7 (11)
Nausea (Gastrointestinal disorders) | 2 (5) | 0 (0) | 6 (9)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 6 (7)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 4 (4)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 5 (5)
Iron Deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (4)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 4 (5)
Toothache (General disorders) | 0 (0) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs are not allowed to publish clinical trial data on their own after trial completion.

DOCUMENTS (2):
  • Study Protocol (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/67/NCT04516967/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/67/NCT04516967/SAP_002.pdf